CLINICAL TRIAL: NCT05165524
Title: Comparison of the Effectiveness of Brightening Creams vs Laser Therapy (QS Nd:YAG 1064nm Laser) in Skin Hyperpigmentation After Sclerotherapy by Objective Measurement: A Randomized Controlled Monocentric Trial
Brief Title: Brightening Cream and Lasers in Post-sclerotherapy Hyperpigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-D0062
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hyperpigmentation; Varicosis
Keywords: laser; Nd:YAG
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser (Active Comparator)
  Interventions: Device: QS Nd:YAG laser
- Cream (Active Comparator)
  Interventions: Drug: Triple cream
- Control (No Intervention)

INTERVENTIONS:
Device: QS Nd:YAG laser — Patients will be treated with Quality-switched (QS) Neodymium-doped yttrium aluminum garnet (Nd:YAG) laser (MedLite® C6) operating at a wavelength of 1064 nm, fluence range from 2.1 J/cm2 to 8.1 J/cm2 with a 4-6mm spot size.
  Arms: Laser
Drug: Triple cream — Patients will be treated with a triple brightening cream (Pigmanorm®), applied daily, three times per week for 12 weeks on the lesion. Interruption for 4 days will be adopted in case of irritation/redness. 50+ sun protection cream will be used as well during the treatment period.
  Arms: Cream

SUMMARY:
The treatment of leg veins and varicosis with sclerotherapy is one of the most frequently performed medical intervention in the western world. The most common local side effects of this treatment are hyperpigmentations caused by hemosiderin deposition in the skin as well as post inflammatory hyperpigmentation.

Although skin hyperpigmentation after sclerotherapy is a common over several months up to years lasting side-effect with a strong aesthetic impact, scanty data exist about treatment options.

Quality-Switched (QS) lasers are efficient in the removal of exogenous and endogenous pigments, such as tattoos as well as epidermal and dermal melanin deposits. The laser light is absorbed by pigment particles, leading to a fragmentation of these particles by a photothermal and photoacoustic effect. Smaller particles can be then phagocyted by macrophages, and transported via the lymphatic system into the lymph nodes. Furthermore, the positive effect of QS lasers in the management of cutaneous siderosis in stasis dermatitis and after sclerotherapy has been described in several cases.

Triple cream including hydroquinone, tretinoin and a topical corticosteroid (eg dexamethasone), is the first line therapy in the treatment of post inflammatory hyperpigmentation.

This randomized controlled study aims to evaluate the efficiency of two well-known depigmentation methods (QS laser and triple cream) for treatment of post sclerotherapy hyperpigmentation, compared with a control group performing no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type I-IV
* Presence of at least 1 postinflammatory hyperpigmentation after sclerotherapy

Exclusion Criteria:

* History of adverse events related to short-pulsed laser therapy
* Pregnant or breast-feeding women
* Intention to become pregnant during the course of the study
* History of intolerance or allergic reaction to triple cream or one of its ingredients
* Prior treatment with parenteral gold therapy
* Inability to understand the study content

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Equivalence of laser and cream in reducing post-sclerotherapy hyperpigmentation as assessed by SHI | 16 weeks
  Equivalence of laser and cream groups in reducing post-sclerotherapy hyperpigmentation as assessed by Skin Hyperpigmentation Index (SHI), ranging from 1 to 4, with higher score indicating a worst hyperpigmentation.

SECONDARY OUTCOMES:
Efficacy of laser and cream in reducing post-sclerotherapy hyperpigmentation compared to control group as assessed by SHI | 4, 8, 12, 16 weeks
  Any reduction of post-sclerotherapy hyperpigmentation in laser and cream compared to control group as assessed by Skin Hyperpigmentation Index (SHI), ranging from 1 to 4, with higher score indicating a worst hyperpigmentation.
Efficacy of laser and cream in reducing post-sclerotherapy hyperpigmentation compared to control group as assessed by PGA | 4, 8, 12, 16 weeks
  Any reduction of post-sclerotherapy hyperpigmentation in laser and cream compared to control group as assessed by 6-point Physician Global Assessment (PGA), based on before-after pictures of lesions assessment, ranging from 1 to 6, with higher scores indicating a better outcome.
Patient's satisfaction related to laser and cream in reducing post-sclerotherapy hyperpigmentation compared to control group | 16 weeks
  Any difference of patient's satisfaction between laser and cream compared to control group as assessed by a 9-point anchored visual analogue scale (VAS), ranging from -4 to +4, with negative scores indicating a worsening of condition, with 0 indicating no difference and with positive scores indicating an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Heidemeyer, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of dermatology, University Hospital Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No